CLINICAL TRIAL: NCT01684423
Title: 30-day, Single-arm Study of the Safety, Efficacy and the Pharmacokinetic and Pharmacodynamic Properties of Oral Rivaroxaban in Children With Various Manifestations of Venous Thrombosis
Brief Title: Oral Rivaroxaban in Children With Venous Thrombosis
Acronym: EINSTEINJunior
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14373; 2011-004539-30 (EudraCT Number)
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Rivaroxaban (BAY59-7939) tablet, OD, Age: 12 - <18 (Experimental): Subjects aged from 12 - <18 years were administered with age and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) IR (immediate-release) tablet once daily (OD) under fed conditions for 30 days. Subjects with a body weight of 14 to less than 50 kilogram (kg) received a dose (equivalent to 20 milligram [mg] in adults) ranging from 5 to 15 mg, and subjects with a body weight (comparable to adults) of greater than or equal to 50 kg received a dose of 20 mg.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Comparator, Age: 12 - <18 years (Active Comparator): Subjects aged from 12 - <18 years received comparator as per standard of care. The dosage given was to be adjusted based on the individual body weight (low molecular weight heparin, fondaparinux) or international normalized ratio (INR) adjusted (vitamin K antagonist).
  Interventions: Drug: Active comparator
- Rivaroxaban (BAY59-7939) tablet, OD, Age: 6 - <12 years (Experimental): Subjects aged from 6 - <12 years were administered with age- and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) IR tablet once daily under fed conditions for 30 days. Subjects with a body weight of 14 to less than 50 kg received a dose (equivalent to 20 mg in adults) ranging from 5 to 15 mg, and subjects with a body weight (comparable to adults) of greater than or equal to 50 kg received a dose of 20 mg.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Rivaroxaban (BAY59-7939) suspension, BID, Age: 6 - <12 years (Experimental): Subjects aged from 6 - <12 years were administered with age- and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) suspension under fed conditions twice daily (BID). Subjects with a body weight of 9 to less than 50 kg received a total daily dose (equivalent to 20 mg in adults) ranging from 6.4 to 15 mg and subjects with a body weight of greater than or equal to 50 kg received a total daily dose of 20 mg.
  Interventions: Drug: Rivaroxaban (BAY59-7939) suspension
- Comparator, Age: 6 - <12 years (Active Comparator): Subjects aged from 6 - <12 years received comparator as per standard of care. The dosage given was to be adjusted based on the individual body weight (low molecular weight heparin, fondaparinux) or INR-adjusted (vitamin K antagonist).
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Subjects were administered with age- and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) IR tablet once daily under fed conditions for 30 days.
  Arms: Rivaroxaban (BAY59-7939) tablet, OD, Age: 12 - <18; Rivaroxaban (BAY59-7939) tablet, OD, Age: 6 - <12 years
Drug: Active comparator — Subjects received comparator as per standard of care. The dosage given was to be adjusted based on the individual body weight (low molecular weight heparin, fondaparinux) or international normalized ratio (INR) adjusted (vitamin K antagonist).
  Arms: Comparator, Age: 12 - <18 years; Comparator, Age: 6 - <12 years
Drug: Rivaroxaban (BAY59-7939) suspension — Subjects aged were administered with age- and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) suspension under fed conditions twice daily.
  Arms: Rivaroxaban (BAY59-7939) suspension, BID, Age: 6 - <12 years

SUMMARY:
The purpose of this study is to find out whether rivaroxaban is safe to use in children and how long it stays in the body. There will also be a check for bleeding and worsening of blood clots.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to < 18 years with documented symptomatic or asymptomatic venous thrombosis treated for at least 2 months or, in case of catheter related thrombosis, treated for at least 6 weeks with LMWH (low molecular weight heparin), , fondaparinux and/or VKA (vitamin K antagonist).
* Informed consent provided and, if applicable, child assent provided

Exclusion Criteria:

* Active bleeding or high risk for bleeding contraindicating anticoagulant therapy
* Symptomatic progression of venous thrombosis during preceding anticoagulant treatment
* Planned invasive procedures, including lumbar puncture and removal of non peripherally placed central lines during study treatment
* An estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
* Hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk or ALT > 5x upper level of normal (ULN) or total bilirubin > 2x ULN with direct bilirubin > 20% of the total
* Platelet count < 50 x 10^9/L
* Hypertension defined as > 95th age percentile
* Life expectancy < 3 months
* Concomitant use of strong inhibitors of both cytochrome P450 isoenzyme 3A4 (CYP3A4) and P-glycoprotein (P-gp), i.e. all human immunodeficiency virus protease inhibitors and the following azole antimycotics agents: ketoconazole, itraconazole, voriconazole, posaconazole, if used systemically
* Concomitant use of strong inducers of CYP3A4, i.e. rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2013-02-19 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (57):
- United States (13):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Orange, California
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - New Hyde Park, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Richmond, Virginia
- Australia (3):
  - Westmead, New South Wales
  - Parkville, Victoria
  - South Brisbane
- Austria (4):
  - Graz, Styria
  - Innsbruck, Tyrol
  - Linz, Upper Austria
  - Vienna
- Canada (5):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Québec
- France (6):
  - Bordeaux
  - Montpellier
  - Nantes
  - Paris
  - Rennes
  - Toulouse
- Germany (6):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Frankfurt am Main, Hesse
  - Dresden, Saxony
  - Lübeck, Schleswig-Holstein
  - Berlin
- Israel (5):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Italy (6):
  - Bari, Apulia
  - Genoa, Liguria
  - Milan, Lombardy
  - Pavia, Lombardy
  - Turin, Piedmont
  - Padua, Veneto
- Netherlands (4):
  - Amsterdam
  - Nijmegen
  - Rotterdam
  - Utrecht
- Switzerland (5):
  - Basel, Canton of Basel-City
  - Sankt Gallen, Canton of St. Gallen
  - Bern
  - Lucerne
  - Zurich

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 10 countries worldwide between 19 February 2013 (first subject first visit) and 01 September 2016 (last subject last visit).
Pre-assignment Details: A total of 68 subjects were screened, of these 4 subjects failed screening. The remaining 64 subjects were randomized, of whom 63 subjects were treated.
Groups:
- Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years: Subjects aged from 12 - <18 years were administered with age and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) IR tablet once daily under fed conditions for 30 days. Subjects with a body weight of 14 to less than 50 kilogram (kg) received a dose (equivalent to 20 milligram [mg] in adults) ranging from 5 to 15 mg, and subjects with a body weight (comparable to adults) of greater than or equal to 50 kg received a dose of 20 mg.
- Comparator, Age: 12 - <18 Years: Subjects aged from 12 - <18 years received comparator as per standard of care.
- Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years: Subjects aged from 6 - <12 years were administered with age- and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) IR tablet once daily under fed conditions for 30 days.
- Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years: Subjects aged from 6 - <12 years were administered with age- and body weight-adjusted oral dose of rivaroxaban (BAY59-7939) suspension under fed conditions twice daily. Subjects with a body weight of 9 to less than 50 kg received a total daily dose (equivalent to 20 mg in adults) ranging from 6.4 to 15 mg and subjects with a body weight of greater than or equal to 50 kg received a total daily dose of 20 mg.
- Comparator, Age: 6 - < 12 Years: Subjects aged from 6 - < 12 years received comparator as per standard of care.
Period: Overall Study
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Comparator, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years | Comparator, Age: 6 - < 12 Years
Started | 11 | 13 | 13 | 19 | 7
Completed | 11 | 13 | 12 | 19 | 7
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Comparator, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years | Comparator, Age: 6 - < 12 Years | Total
Number analyzed (Participants) | 11 | 13 | 13 | 19 | 7 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.5 (1.2) | 14.8 (1.0) | 8.5 (2.1) | 8.3 (1.9) | 9.0 (2.0) | 11.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 5 | 6 | 3 | 29
  Male | 3 | 6 | 8 | 13 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Major and Clinically Relevant Non-Major Bleeding Events
Description: Central independent adjudication committee (CIAC) classified bleeding as follows: Major bleeding is defined as overt bleeding and:
  * associated with a fall in hemoglobin of 2 gram/decilitre (g/dL) or more, or
  * leading to a transfusion of the equivalent of 2 or more units of packed red blood cells or whole blood in adults, or
  * occurring in a critical site, e.g. intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal, or
  * contributing to death.
  Clinically relevant non-major bleeding is defined as overt bleeding not meeting the criteria for major bleeding, but associated with:
  * medical intervention, or
  * unscheduled contact (visit or telephone call) with a physician, or
  * cessation (temporary) of study treatment, or
  * discomfort for the child such as pain or
  * impairment of activities of daily life (such as loss of school days or hospitalization).
Time Frame: From start of study drug administration until end of the 30-day treatment period
Population: Full analysis set. Data was evaluated only for subjects who received active study medication.
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Comparator, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years | Comparator, Age: 6 - < 12 Years
Number analyzed (Participants) | 11 | 13 | 13 | 19 | 7
Participants
  Major bleeding events | 0 | 0 | 0 | 0 | 0
  Clinically relevant non-major bleeding events | 3 | 0 | 0 | 1 | 0

2. Secondary Outcome: Number of Subjects With Symptomatic Recurrent Venous Thromboembolism
Description: The occurrence of recurrent venous thromboembolism was summarized by age group. Symptomatic recurrence of venous thrombosis was documented by the appropriate imaging test.
Time Frame: From start of study drug administration until end of the 30-day treatment period
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Comparator, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years | Comparator, Age: 6 - < 12 Years
Number analyzed (Participants) | 11 | 13 | 13 | 19 | 7
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Subjects With Asymptomatic Deterioration in Thrombotic Burden
Description: The occurrence of asymptomatic deterioration in thrombotic burden was summarized by age group. Asymptomatic deterioration in thrombotic burden was documented by the appropriate imaging test and the results were classified as normalized, improved, no relevant change, deteriorated, not evaluable or not available.
Time Frame: Repeat imaging at the end of the 30 day treatment period
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Comparator, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years | Comparator, Age: 6 - < 12 Years
Number analyzed (Participants) | 11 | 13 | 13 | 19 | 7
Participants
  Normalized | 3 | 2 | 2 | 4 | 1
  Improved | 4 | 0 | 8 | 9 | 4
  No relevant change | 0 | 0 | 1 | 2 | 0
  Deteriorated | 0 | 0 | 0 | 0 | 0
  Not evaluable | 0 | 2 | 0 | 0 | 1
  Not available | 4 | 9 | 2 | 4 | 1

4. Secondary Outcome: Change From Baseline in Prothrombin Time at Specified Time Points
Description: Prothrombin time is a global clotting test used for the assessment of the extrinsic pathway of the blood coagulation cascade.
Time Frame: 0 hours (pre-dose) to 8 hours post-dose on Day 15 and 24 hours post-dose on Day 31
Population: Pharmacodynamic analysis set (N=42) included all subjects with at least one blood sample for clotting parameters in accordance with the pharmacodynamic sampling strategy.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years
Number analyzed (Participants) | 11 | 12 | 19
seconds
  Day 15: 2 to 4 hours post-dose | 8.964 (3.822) | 9.083 (2.513) | 3.147 (2.099)
  Day 15: 6 to 8 hours post-dose | 4.218 (2.977) | 2.817 (1.628) | 1.984 (1.341)
  Day 31: 10 to 16 hours post-dose | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | 0.156 (1.155)
  Day 31: 20 to 24 hours post-dose | -0.082 (1.020) | -0.327 (1.332) | NA (NA) — Data is not available because no subjects were evaluated for the given time points.

5. Secondary Outcome: Change From Baseline in Activated Partial Thromboplastin Time at Specified Time Points
Description: The Activated partial thromboplastin time (aPTT) is a screening test for the intrinsic pathway.
Time Frame: 0 hours (pre-dose) to 8 hours post-dose on Day 15 and 24 hours post-dose on Day 31
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years
Number analyzed (Participants) | 11 | 12 | 19
seconds
  Day 15: 2 to 4 hours post-dose | 10.982 (4.470) | 12.818 (5.210) | 2.995 (5.616)
  Day 15: 6 to 8 hours post-dose | 6.136 (2.641) | 5.900 (4.942) | 1.858 (4.774)
  Day 31: 10 to 16 hours post-dose | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | -0.483 (6.488)
  Day 31: 20 to 24 hours post-dose | 1.345 (3.190) | 1.240 (4.992) | NA (NA) — Data is not available because no subjects were evaluated for the given time points.

6. Secondary Outcome: Anti-factor Xa Values at Specified Time Points
Description: The individual anti-Factor Xa activity was determined ex-vivo using a photometric method.
Time Frame: 0 hours (pre-dose) to 8 hours post-dose on Day 15 and 24 hours post-dose on Day 31
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years
Number analyzed (Participants) | 11 | 12 | 19
microgram per liter (mcg/L)
  Day 15: pre-dose | 16.081 (6.136) | 8.136 (3.069) | 31.553 (25.416)
  Day 15: 2 to 4 hours post-dose | 185.481 (53.326) | 252.853 (71.072) | 99.415 (54.415)
  Day 15: 6 to 8 hours post-dose | 105.223 (54.339) | 68.670 (32.845) | 77.929 (50.074)
  Day 31: 10 to 16 hours post-dose | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | 30.927 (18.037)
  Day 31: 20 to 24 hours post-dose | 16.038 (7.653) | 8.409 (3.664) | NA (NA) — Data is not available because no subjects were evaluated for the given time points.

7. Secondary Outcome: Concentration of Rivaroxaban in Plasma as a Measure of Pharmacokinetics at Specified Time Points
Description: Geometric and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: 0 hours (pre-dose) to 8 hours post-dose on Day 15 and 24 hours post-dose on Day 31
Population: Pharmacokinetic analysis set (N= 42) included all subjects with at least one pharmacokinetic sample in accordance with the pharmacokinetic sampling strategy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years
Number analyzed (Participants) | 11 | 12 | 19
microgram per liter (mcg/L)
  Day 15: pre-dose | 20.4822 (40.6726) | 7.4367 (152.9768) | 41.6025 (183.6873)
  Day 15: 2 to 4 hours post-dose | 219.6933 (35.7518) | 240.6319 (18.3387) | 119.2201 (52.9889)
  Day 15: 6 to 8 hours post-dose | 124.6723 (49.1882) | 96.8051 (41.8155) | 100.5992 (52.6497)
  Day 31: 10 to 16 hours post-dose | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | NA (NA) — Data is not available because no subjects were evaluated for the given time points. | 43.5223 (81.7283)
  Day 31: 20 to 24 hours post-dose | 21.3252 (43.1274) | 9.4654 (167.7545) | NA (NA) — Data is not available because no subjects were evaluated for the given time points.

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 day post study treatment
Arm/Group | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years | Comparator, Age: 12 - <18 Years | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years | Comparator, Age: 6 - < 12 Years
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/13 | 0/13 | 2/19 | 0/7
Other Adverse Events (participants affected / at risk) | 9/11 | 8/13 | 6/13 | 12/19 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years (N=11) | Comparator, Age: 12 - <18 Years (N=13) | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years (N=13) | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years (N=19) | Comparator, Age: 6 - < 12 Years (N=7)
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Influenza B virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 12 - <18 Years (N=11) | Comparator, Age: 12 - <18 Years (N=13) | Rivaroxaban (BAY59-7939) Tablet, OD, Age: 6 - <12 Years (N=13) | Rivaroxaban (BAY59-7939) Suspension, BID, Age: 6 - <12 Years (N=19) | Comparator, Age: 6 - < 12 Years (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days